CLINICAL TRIAL: NCT01812057
Title: Dexamethasone as an Analgesic Adjunct for Post-cesarean Delivery Pain Relief
Brief Title: Dexamethasone for Post-cesarean Delivery Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00041334
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
Keywords: Anesthesia; Cesarean Section; Pain, Postoperative; Postoperative Nausea and Vomiting; Dexamethasone; Injections, Spinal; morphine
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 8 mg IV given intraoperatively as a one-time dose.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Sodium chloride 0.9% (5 ml) given IV intraoperatively as a one time dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8 mg IV (as a one time dose)
  Arms: Dexamethasone
Drug: Placebo — Sodium Chloride 0.9% -5 ml
  Other Names: Sodium Chloride 0.9%
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare post-cesarean section consumption of pain medication between two groups of patients undergoing scheduled cesarean section at term gestation who receive a single-dose of intraoperative steroid (dexamethasone 8 milligrams) versus placebo at 24 hours after surgery. The hypothesis is that a single perioperative dose of dexamethasone 8 mg will significantly reduce postoperative opioid consumption at 24 h in women having cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
Steroids have been used to reduce inflammation and tissue damage in a variety of conditions, have potent immunomodulatory effects, and are a mainstay in the treatment of acute allograft rejection. Dexamethasone has been shown to be a safe and effective anti-emetic therapy for patients undergoing cesarean section surgery with spinal anesthesia containing morphine.

However, recent evidence suggests that dexamethasone may also play a role in reducing post-operative pain and opioid consumption. Early studies in patients undergoing dental procedures showed that glucocorticoids were effective in reducing postoperative pain and edema. Multiple recent studies have also investigated the potential analgesic benefit of a single perioperative dose of dexamethasone, but the results have been inconsistent. The effect of single-dose, intraoperative, intravenous dexamethasone therapy on post-operative pain and opioid consumption has not yet been studied in patients undergoing cesarean section.

Pain is a significant source of morbidity for many women following cesarean section, and has serious consequences beyond the immediate post-operative period. Patients with poorly-controlled pain may have difficulty with ambulation that can lead to atelectasis, pneumonia, and venous thromboembolism.

Poor maternal pain control may also affect the infant by interfering with bonding and breastfeeding. Reduction of post-operative opioid consumption is desirable because it may also reduce the incidence of opioid-induced side effects such as sedation, constipation, nausea, vomiting and pruritus. Some evidence suggests that the severity of post-operative pain following cesarean section may predict progression to chronic pain, and postpartum depression.

Although 10 to 18% of women who undergo cesarean section will experience chronic pain following surgery, it is difficult to predict those patients who will experience this complication. Recent investigations have shown that patient responses to standardized painful stimuli prior to surgery help predict severity of post-operative pain and possibly progression to chronic pain. This type of information could potentially help to tailor the clinical management of patients at risk for severe and/or chronic post-operative pain to improve outcomes for these patients. Landau and colleagues have described a simple and minimally-invasive method of assessing response to noxious stimuli using a von-Frey filament to obtain a mechanical temporal summation score.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class 1, 2 and 3
* Gestational age > 37 weeks
* scheduled for elective cesarean delivery
* spinal or combined spinal epidural anesthesia
* 18 years or older
* speak English

Exclusion Criteria:

* BMI > 45 kg/m2
* Diabetes Mellitus (Type 1, 2 and gestational)
* mild or severe preeclampsia
* history of intravenous drug or opioid abuse
* previous history of chronic pain syndrome
* history of opioid use in the past week
* receipt of an antiemetic within 24 h prior to surgery
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-12; Primary Completion 2016-05-27 (Actual); Study Completion 2016-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Allen, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 52 subjects that were enrolled, 3 subjects were not randomized due to later being deemed ineligible for the study; therefore, 49 subjects started on study.
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 25 | 24
Completed | 23 | 24
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (4.7) | 30.63 (5.71) | 31.40 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 17 | 14 | 31
  Race/Ethnicity: Black/African American | 6 | 5 | 11
  Race/Ethnicity: Asian/Indian | 0 | 3 | 3
  Race/Ethnicity: Hispanic | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption at 24 Hours Post-op
Description: The primary outcome will be the cumulative morphine consumption at 24 h in the two study groups. All postoperative opioids were converted to IV morphine equivalents using the following conversion factors: 100 micrograms IV = 10 mg IV morphine, 20 mg oxycodone po = 10 mg IV Morphine
Time Frame: 24 hours from admission to Postanesthesia care unit (PACU)
Measure: Median (Inter-Quartile Range); unit: milligram
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
milligram | 15 [7.5 to 20.0] | 13.75 [2.5 to 31.25]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.740, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Scores Between the Groups at 2 Hours.
Description: Pain scores were measured using a numeric rating scale with a range from 0 to 10, with 0 meaning no pain and 10 indicating the most severe pain.
Time Frame: 2 hours from admission to postanesthesia care unit (PACU)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale
  Pain Score at rest | 2 [0.0 to 4.0] | 3.5 [1.5 to 5.0]
  Pain Score with movement | 5 [2.0 to 7.0] | 5 [4.0 to 7.0]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Pain Score at rest at 2 hours; p = 0.171, t-test, 2 sided
Statistical Analysis 2: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Pain Score with movement at 2 hours; p = 0.204, t-test, 2 sided

3. Secondary Outcome: Time to Administration of First Rescue Analgesic Request Between the Groups.
Description: Time in minutes from admission to PACU to the first request by the patient for oral oxycodone (analgesia) administration for pain
Time Frame: PACU admission to discharge from PACU an average of 2 hours
Population: Analysis was based on all 47 patients who completed the study.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
minutes | 52.5 [22.5 to 88.5] | 70 [30 to 112]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.1965, Log Rank

4. Secondary Outcome: Cumulative Opioid Consumption at 48 Hours Between the Groups
Description: The secondary outcome was the cumulative morphine consumption at 48 h in the two study groups. All postoperative opioids were converted to IV morphine equivalents using the following conversion factors: 100 micrograms IV = 10 mg IV morphine, 20 mg oxycodone po = 10 mg IV Morphine
Time Frame: Admission to PACU through 48 hours
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
milligrams | 20 [10.0 to 40.0] | 22.5 [3.75 to 48.75]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.709, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Pain Scores Between the Groups at 24 Hours.
Description: as for outcome 2
Time Frame: 24 hours from PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale
  Pain Score at rest | 2 [0.0 to 3.0] | 2.5 [1.0 to 4.25]
  Pain Score with movement | 5 [3.0 to 7.0] | 5 [4.0 to 6.75]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Pain Score at rest at 24 hours; p = 0.267, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Pain Score with movement at 24 hours; p = 0.518, t-test, 2 sided

6. Secondary Outcome: Pain Scores Between the Groups at 48 Hours.
Description: as for outcome 2
Time Frame: 48 hours from PACU Admission
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale
  Pain Score at rest | 2.0 [0.0 to 3.0] | 2.0 [0.0 to 4.0]
  Pain Score with movement | 4.0 [3.0 to 6.0] | 5.0 [3.0 to 7.0]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Pain Score at rest at 48 hours; p = 0.491, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Pain Scores with movement at 48 hours; p = 0.525, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Cumulative Opioid Consumption at 24 Hours Between MTS Groups
Description: Mechanical temporal summation (MTS) was assessed using A 180 g Von Frey Filament was applied to the volar aspect of the dominant forearm, and subjects were asked to rate pain scores (NRS 0-100, 0 = no pain and 100= worst pain possible) after the 1st and 11th tap. A difference < 1 was recorded as MTS negative, and a difference > or = 1 was recorded as MTS positive.
Time Frame: 24 hours from admission to Postanesthesia care unit (PACU)
Population: Analysis was based on all 47 patients who completed the study.
Measure: Median (Inter-Quartile Range); unit: milligrams
Groups:
- Positive MTS Score: Positive MTS score is defined as change of >1 in MTS score between 1st tap and 11th tap of 180 gram von Frey filament.
- Negative MTS Score: Negative MTS score is defines as change of less than or equal to 1 in MTS scores between 1st tap and 11th tap.
Arm/Group | Positive MTS Score | Negative MTS Score
Number analyzed (Participants) | 9 | 38
milligrams | 17.5 [7.5 to 32.5] | 15 [2.5 to 25]
Statistical Analysis 1: Comparison: Positive MTS Score vs Negative MTS Score; Test type: Superiority; p = 0.355, Wilcoxon (Mann-Whitney); Total opioid consumption at 24 hours; We also performed a multivariable regression analysis to determine factors associated with 24h opioid consumption accounting for MTS category, demographic factors, study group allocation (dexamethasone vs placebo) and a preoperative questions to assess patients anxiety, anticipated pain scores after surgery and anticipated analgesic need after surgery. At each step of backward variable selection, we eliminate the factor with the largest p-value over 0.05.In the final model MTS was not associated with 24h opioid consumption parameter estimate (standard error) = 9.15 (5.27), p=0.09

8. Secondary Outcome: Incidence of Chronic Persistent Pain at 8 Weeks
Description: Patients answered a questionnaire at 8 weeks to determine whether they still had persistent surgical site pain 8 weeks following surgery
Time Frame: 8 weeks from the day of surgery
Population: Analysis was based on available data from both arms including 26 patients. Data was missing for 13 patients in dexamethasone group and 8 patients in placebo group.
Measure: Count of Participants; unit: Participants
Groups:
- Dexamethasone: Dexamethasone 8 mg IV given intraoperatively as a one-time dose. ...
- Placebo: Sodium chloride 0.9% (5 ml) given IV intraoperatively as a one time dose. ...
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 10 | 16
Participants | 2 | 6
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.420, Fisher Exact; Chronic pain at 8 weeks

9. Secondary Outcome: Incidence of Chronic Persistent Pain at 6 Months
Description: Patients answered a questionnaire at 6 months to determine whether they still had persistent surgical site pain 6 months following surgery
Time Frame: 6 months from the day of surgery
Population: Analysis was based on available data from both arms including 25 patients. Data was missing for 11 patients in dexamethasone group and 11 patients in placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 3 | 1
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.322, Fisher Exact

10. Secondary Outcome: Pain Scores Between MTS Groups
Description: Mechanical temporal summation (MTS) was assessed using A 180 g Von Frey Filament was applied to the volar aspect of the dominant forearm, and subjects were asked to rate pain scores (NRS 0-100, 0=no pain and 100=worst pain possible) after the 1st and 11th tap. A difference < 1 was recorded as MTS negative, and a difference > or = 1 was recorded as MTS positive.
Time Frame: 24 hours after PACU admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Positive MTS Score | Negative MTS Score
Number analyzed (Participants) | 9 | 38
units on a scale
  Pain scores at rest at 24 hours | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 4.0]
  Pains scores on movement at 24 hours | 5.0 [3.0 to 7.0] | 4.0 [4.0 to 6.0]
Statistical Analysis 1: Comparison: Positive MTS Score vs Negative MTS Score; 24 hour pain scores at rest between MTS groups; Test type: Superiority; p = 0.805, Wilcoxon (Mann-Whitney); We also performed a multivariable regression analysis to determine factors associated with Pain scores at rest at 24 hours accounting for MTS category, demographic factors, study group allocation (dexamethasone vs placebo) and a preoperative questions to assess patients anxiety, anticipated pain scores after surgery and anticipated analgesic need after surgery. At each step of backward variable selection, we eliminate the factors with the largest p-value over 0.05. MTS category was not included in the final model for 24 h pain scores at rest
Statistical Analysis 2: Comparison: Positive MTS Score vs Negative MTS Score; Pain scores on movement at 24h; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney); We also performed a multivariable regression analysis to determine factors associated with Pain scores at rest at 24 hours accounting for MTS category, demographic factors, study group allocation (dexamethasone vs placebo) and a preoperative questions to assess patients anxiety, anticipated pain scores after surgery and anticipated analgesic need after surgery. At each step of backward variable selection, we eliminated the factors with the largest p-value over 0.05. MTS category was not included in the final model for 24 h pain scores on movement

11. Secondary Outcome: Incidence of Intraoperative Nausea and Vomiting (IONV) and Need for Rescue Antiemetics.
Description: Incidence of intraoperative nausea and vomiting and need for rescue antiemetics were recorded during surgery. Patient who reported a nausea score on a 11 point NRS where 0=no nausea and 10 = the worse nausea possible. Patients who retched or vomited were reported to have vomited. Patients receiving any antiemetic during surgery were recorded as those requesting ( needing) rescue antiemetic.
Time Frame: From spinal anesthesia placement to end of surgery, approximately 70 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
Participants
  Incidence of intraoperative nausea | 5 | 2
  Intraoperative need for rescue antiemetic | 10 | 9
  Incidence of intraoperative vomiting | 4 | 5
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority — Intraoperative nausea and vomiting; p = 0.245, Fisher Exact
Statistical Analysis 2: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.676, Chi-squared; Need for intraoperative antiemetics
Statistical Analysis 3: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

12. Secondary Outcome: Incidence of Intraoperative Pruritus
Description: pruritus was defined as patients reporting a pruritus score of greater than o on a numerical rating scale with o=no pruritus and 10= worst pruritus
Time Frame: From spinal anesthesia placement to end of surgery, approximately 70 minutes
Population: No data was collected on intraoperative pruritus on any participants.
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Incidence of Postoperative Pruritus
Description: Incidence of postoperative pruritus was calculated based on their postoperative pruritus scores measured at 2 hours, 24 hours and 48 hours. Median of the scores recorded at three time points was calculated.
  If median score >0 then patient experienced postoperative pruritus.
Time Frame: 48 hours from admission to PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
Participants | 16 | 17
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.924, Chi-squared; Incidence of postoperative pruritus

14. Secondary Outcome: Need for Intraoperative Analgesic Supplementation
Description: Need for intraoperative analgesic supplementation was determined by patients who required intraoperative analgesics for pain
Time Frame: From spinal anesthesia placement to end of surgery, approximately 70 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
Participants | 4 | 3
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.700, Fisher Exact

15. Secondary Outcome: Incidence of Post-operative Nausea and Vomiting (PONV) and Need for Rescue Antiemetics
Description: Patients who had experienced Postoperative nausea either reported postoperative nausea scores at 2, 24 and 48 hours from >0, reported an episode of vomiting or received an antiemetic were recorded as experiencing PONV.
  Patients who received at least one rescue antiemetic postoperatively were recorded as requiring a rescue antiemetic
Time Frame: 2, 24 and 48 hours from PACU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
Participants
  Incidence of PONV at 24 hours | 9 | 13
  Postoperative need for rescue antiemetics | 10 | 18
  Incidence of PONV at 48 hours | 1 | 2
  Incidence of PONV at 2 h | 9 | 14
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.302, Chi-squared; Incidence of PONV at 24 h
Statistical Analysis 2: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.028, Chi-squared; Postoperative need for rescue antiemetic
Statistical Analysis 3: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.188, Chi-squared

16. Secondary Outcome: Incidence of Wound Complications
Description: Patients were assessed for signs of surgical wound inspection by the obstetric team following surgery
Time Frame: 24 hours from PACU admission
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 23 | 24
Participants | 0 | 0

17. Secondary Outcome: Blood Pressure Measurements Obtained by the Standard of Care Non-invasive Blood Pressure Monitor Compared With the Continuous Noninvasive Arterial Pressure (CNAP)
Time Frame: Intraoperatively
Population: No data was collected intraoperatively using CNAP on any participants.
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time PACU admission until 48 hours from PACU admission.
Description: Adverse Event reporting for this study were limited to surgical site infections and wound dehiscence assessed by the obstetricians daily
Arm/Group | Dexamethasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

LIMITATIONS AND CAVEATS:
The study was ended prior to completion of total planned enrollment of 104 subjects due to a change in clinical practice regarding post-operative pain medications that would have confounded the results of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes